CLINICAL TRIAL: NCT07186829
Title: Randomised Controlled Evaluation of the Repair of Extra-articular Fractures of the Metacarpals and First Phalanges of the Long Fingers: Centromedullary Screw Osteosynthesis Versus Pinning Versus Locked Plate.
Brief Title: Randomised Controlled Evaluation of the Repair of Extra-articular Fractures of the Metacarpals and First Phalanges of the Long Fingers
Acronym: FinXger
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL24_0382
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hand Fractures
Keywords: hand; fracture; ostheosynthesis; screw; plate; k-wire; phalanx; metacarpal
MeSH Terms: conditions — Fractures, Bone | interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Percutanous pinning (Active Comparator): closed reduction, two percutaneous pins
  Interventions: Device: Percutanous pinning
- Locked plate (Active Comparator): open reduction, dorsal approach, 3 screws proximal and distal
  Interventions: Device: Locked plate
- Intramedullary screw (Active Comparator): 1 cm dorsal incision, closed reduction, internal compression screw
  Interventions: Device: Intramedullary screw

INTERVENTIONS:
Device: Percutanous pinning — Similar to arm - closed reduction, two percutaneous pins
  Other Names: K-wire; Kirchner wire
  Arms: Percutanous pinning
Device: Locked plate — Similar to arm - open reduction, dorsal approach, 3 screws proximal and distal
  Other Names: Locking plate
  Arms: Locked plate
Device: Intramedullary screw — Similar to arm - 1 cm dorsal incision, closed reduction, internal compression screw
  Other Names: Intramedullary compression screw; Herbert screw
  Arms: Intramedullary screw

SUMMARY:
The goal of this randomized controlled trial is to compare the effectiveness, complications, and cost-effectiveness of three surgical techniques (intramedullary screw fixation, locked plating, and percutaneous pinning) for treating simple transverse extra-articular fractures of the proximal phalanges and metacarpals (excluding the thumb) in adult patients. The main questions it aims to answer are:

The primary outcome is to define which technique results in better functional outcomes, as measured by pulp-to-palm distance at 6 weeks?

The main secondary outcome is to define which technique has lower complication rates and is more cost-effective over 12 months?

Participants will be randomly assigned to one of the three surgical techniques (intramedullary screw fixation, locked plating, or percutaneous pinning). Follow-up visits at weeks: 3, 6 and months: 3,6 and final follow-up at 12 months will assess hand function, range of motion, grip strength, radiographic healing, complications, satisfaction, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Simple transverse extra-articular fractures of proximal or diaphyseal phalanges/metacarpals with surgical indication

Exclusion Criteria:

* Thumb fracture, open fracture, ischemia, pathological fracture, previous fracture, denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Pulp-to-palm distance at 6 weeks | at 6 weeks
  Global range of motion measured by pulp-to-palm distance at 6 weeks

SECONDARY OUTCOMES:
Range of motion | at 3 weeks, 6 weeks, 3months, 6 months and 12 months
  Flexion and extension angle in degrees for MCP and PIP joints
Bone Healing | 3weeks, 6 weeks, 3months, 6months, 12months
  Radiographical bone healing with routine AP and lateral x-rays
Cost analysis of each technique at 12months | 12months
  Relative cost between each technique for intra and post operative care
Complications | 3weeks, 6 weeks, 3months, 6months, 12months
  Every clinical and paraclinical complication that may occur
Grip strength | 3months, 6months, 12months
  Grip strength measured in kg with a validated JAMAR® Hand Dynamometer
QuickDASH PROM score | 3months, 6months, 12months
  Functionnal recovery evaluated with the QuickDASH PROM score
Patient satisfaction | 3months, 6months, 12months
  Patient satisfaction evaluated with visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Emmanuel Chammas, MD, MSc, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No